CLINICAL TRIAL: NCT03798171
Title: Reduction of Exit Site Infection in Peritoneal Dialysis Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, Department of nephrology, Tel-Aviv Sourasky Medical Center
Other Study IDs: 0077-18-TLV
Record Dates: First submitted 2019-01-07; First posted 2019-01-09 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Peritoneal Dialysis Catheter Infection
Keywords: peritoneal dialysis; exit site; infection; peritonitis
MeSH Terms: conditions — Infections; Peritonitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In peritoneal dialysis patients, the presence of the catheter presents a risk of infection - exit site infection, tunnel infection or peritonitis. In our dialysis unit, we noticed a rise in exit-site infection associated with organisms derived from contaminated water. Therefore we decided to change the exit-site care in our unit.

This is a prospective observational single center study, that compares exit-site infection rated in peritoneal dialysis patients before and after our policy change for exit-site care.

DETAILED DESCRIPTION:
Peritoneal dialysis is a method for renal replacement therapy that uses the peritoneal membrane for exchange of fluids and dissolved substance . A catheter is surgically inserted with one end in the abdomen and the other protruding from the skin, in order to allow fluid exchange.

The presence of the catheter presents a risk of infection - exit site infection, tunnel infection or peritonitis - a cause of morbidity and treatment failure.

Infection prevention is based, among other measures, on aseptic handeling of catheter exit-site. In our dialysis unit, we noticed a rise in pseudomonas exit-site infection and other organisms associated with contaminated water. Therefore we decided to change the exit-site care in our unit. Similar to central catheters handeling, we decided to cover the catheter exit-site during water exposure, and to change the prophylactic exit-site antibiotic regimen.

This is a prospective observational single center study. All peritoneal dialysis patients in our institue will be counseled about change in exit-site care. For prevention of water exposure the patients will use stoma bags around the catheter during showers. After the shower, the exit-site is cleaned with a chlorhexidine based solution, an antibiotic cream is applied (Mupirocin) and dressed with a clean gauze.

The patients will be followed for 3 years for adverse events. The number of infectious episodes will be recorded and compared to historical data (January 2015-December 2017).

ELIGIBILITY:
Inclusion Criteria:

* peritoneal dialysis patients capable to sign an informed consent or have an official guardian

Exclusion Criteria:

* patient's refusal

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: peritoneal dialysis patients in Tel Aviv Sourasky medical center
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-05-15 (Actual); Primary Completion 2021-05-15 (Estimated); Study Completion 2021-05-15 (Estimated)

PRIMARY OUTCOMES:
exit-site infection rate | 36 months
  number of exit-site infection during 3 years of follow up, compared to historical data

SECONDARY OUTCOMES:
peritonitis rate | 36 months
  number of peritonitis episodes during 3 years of follow up, compared to historical data

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical Canter, Tel Aviv, Israel